CLINICAL TRIAL: NCT01761903
Title: Functional Connectivity of the Basal Ganglia in Primary Focal Dystonia
Brief Title: Functional Connectivity in Primary Focal Dystonia
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0289
Record Dates: First submitted 2012-12-06; First posted 2013-01-07 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Focal Dystonia: Volunteers with primary focal dystonia
- Healthy Controls: 'Healthy' volunteers, consisting of people of the same age as the PFD volunteers, w/o a diagnosis of PFD.

SUMMARY:
In this study we are looking at primary focal dystonias, including dystonias of the limbs, eyes, jaw or face, neck, and vocal chords. This study will use magnet resonance imaging (MRI) to see how the brain reacts while resting and doing a finger-tapping task.

The investigators will test the hypothesis that disturbances in functional connectivity within the motor, affective and cognitive basal ganglia networks in primary focal dystonia (PFD) underlie the motor and non-motor symptoms in this disorder.

DETAILED DESCRIPTION:
After written consent is obtained, all subjects undergo a neurological examination by a board certified neurologist and complete a Montreal Cognitive Assessment and Edinburgh Handedness Inventory. Primary focal dystonia (PFD) patients will have their dystonia assessed with commonly used clinical rating scales for dystonia using Unified Dystonia Rating Scale,Fahn-Marsden Scale, Global Dystonia Rating Scale, Toronto Western Spasmodic Torticollis Rating Scale-TWSTRS,and the Jankovic Rating Scale for blepharospasm. Patients and controls will have affective symptoms assessed using the Liebowitz Social Anxiety Scale, Hospital Anxiety and Depression Scale,Yale-Brown Obsessive Compulsive Scale,and Beck Depression Inventory. Clinical evaluations will be performed at the University of Colorado Denver and Denver Veterans Affairs (VA) Hospital Brain Imaging Center on the Anschutz Medical Campus, prior to Magnetic Resonance Imaging (MRI) scanning. Consenting, exam, and clinical scale assessments are estimated to take 30-40 minutes to complete.

MRI scanning protocol

MRI scanning will be performed using an 8-channel head coil and a 3 Tesla General Electric (GE) Signa MR scanner system that is FDA-approved for clinical MR scanning. The principal investigator and/or a co-investigator will be present for every scanning session. Head motion will be minimized using cushions and passive restraints. The total MRI scanning session will take approximately 50-60 minutes, including set-up time and scan time, and includes the following MRI runs:

1. Anatomic scans: A high-resolution 3D spoiled gradient echo T1-weighted image (~8 minutes) will be collected for image registration and normalization. The subject simply rests while the sequence is run. A diffusion tensor imaging (DTI) scan (~10 minutes) will be acquired using a double spin-echo diffusion echo-planar imaging (EPI) sequence and 32 diffusion directions.
2. Resting-state task (~6 min): Subject remains motionless with eyes closed and tries not to sleep or think of anything in particular.
3. Motor tapping task (~6 min): Subject performs a sequential five-finger finger-tapping sequence in 30 sec blocks that alternate with 30 sec of rest. The tapping task was designed to minimize variance in performance between and within individuals and so is paced with an audible cue. During the rest condition the subject is to remain motionless and not think of anything in particular. A similar motor task has been shown to be feasible in primary dystonia (PD) patients and lead to striatal dopamine release.
4. Repeat of motor task functional Magnetic Resonance Imagine (fMRI) scan (~6 minutes) - subject uses opposite hand to perform sequential finger tapping task, but otherwise scan is identical to above.

Behavioral assessments

1. Button presses during finger-tapping task scanning will be recorded using an MRI-compatible five-button response unit.
2. Surface electromyographic (EMG) recordings will be obtained during resting-state and motor task fMRI scans to assess spontaneous dystonic motor activity, movement during rest, and muscle activity during tapping. Simultaneous EMG monitoring will be performed using a EMG Amplifier designed for fMRI acquisition and small adhesive pad EMG electrodes taped to the skin.

ELIGIBILITY:
Inclusion Criteria:

* English as their primary language
* Volunteers with PFD and healthy controls
* PFD volunteers must be on a stable dose of all dystonia and neuroactive drugs (e.g. antidepressants) for one month prior to enrollment
* PFD volunteers must not have been injected with botulinum toxin within the prior 2 months

Exclusion Criteria:

* Any contraindication to MRI scanning
* Any untreated neurological or psychiatric condition
* Evidence on neurological exam of any potentially confounding neurological disorder (e.g., Parkinson disease, Essential Tremor, etc.)
* Evidence of significant cognitive impairment (all subjects assessed using the Montreal Cognitive Assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult-onset primary focal dystonia patients 18 years old and older with symptoms affecting muscles of the eye (blepharospasm), jaw or face (cranial), neck (cervical), limbs (arm/leg), or vocal chords.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Contrast between Primary Focal Dystonia (PFD) and Healthy Controls (HC) | Day 1
  Primary outcome measures for the first aim is a second level contrast between Primary Focal Dystonia (PFD) and Healthy Controls (HC) of the statistical parametric maps of correlation coefficients (measures of functional connectivity associated with predefined basal ganglia regions of interest) at rest and during a tapping motor task.
Correlation between basal ganglia motor network functional connectivity measures and total PFD clinical assessment scale scores | Day 1
  The primary outcome measure for the second aim is the strength of correlation between basal ganglia motor network functional connectivity measures and total PFD clinical assessment scale scores.

SECONDARY OUTCOMES:
Evaluation of Lateralization | Day 1
  Secondary outcome measures will include within group comparisons of statistical parametric maps of correlation coefficients to investigate lateralization (left versus right side of onset; left versus right tapping hand).
Statistical dependence between symptoms and measures of basal ganglia functional connectivity | Day 1
  Secondary outcome measures will include measuring statistical dependence between symptoms (assessment by clinical scale scores) and measures of basal ganglia functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States